CLINICAL TRIAL: NCT05941637
Title: An Expanded Access Program to Axitinib is Available for Patients With Advanced Forms of Kidney Cancer (Ductal; Papillary; Chromophobic; Oncocytic), Confirmed Mutations in VHL, PBRM1 / BAP1, SETD2, VEGF), for Whom Standard Systemic Therapy Has Failed or Progressed, in Whom There Are no Satisfactory Treatment Alternatives and Who Are Not Eligible for Other Clinical Trials.
Brief Title: An Expanded Access Program to Axitinib is Available for Patients With Advanced Forms of Kidney Cancer (Ductal; Papillary; Chromophobic; Oncocytic) With Mutations in VHL, PBRM1 / BAP1, SETD2, VEGF)
Status: No longer available | Type: Expanded Access
Sponsor: Lynkcell Europe (Other)
Responsible Party: Sponsor
Other Study IDs: EAR688789-CH
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Clear Cell Kidney Cancer; Kidney Cancer; Kidney Cancer With PBRM1/BAP1/VHL/SETD2 Mutations
MeSH Terms: conditions — Kidney Neoplasms | interventions — Axitinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Axitinib 5 MG — Patients will receive Axitinib (AG 013736) is a multi-target inhibitor of VEGFR1, VEGFR2, VEGFR3, PDGFRβ, and c-Kit - 5mg daily
  Other Names: INLYTA; AG-013736

SUMMARY:
Kidney cancer belongs to a heterogeneous group of tumors and is the most common oncourological disease; up to 80% of cases are clear cell carcinoma.

DETAILED DESCRIPTION:
The study of rare hereditary forms of clear cell kidney cancer (CRP) made it possible to identify the VHL gene, germline mutations which lead to the development of the Hippel-Lindau syndrome, and somatic mutations are characteristic of sporadic CRP. The second most frequent mutation independent of VHLmut is the PBRM1 gene involved in chromatin remodeling. PBRM1 mutations are positively correlated with SETD2 mutations and negatively correlated with BAP1 mutations. Depending on the status of PBRM1/BAP1 mutations, tumors are characterized by different pathomorphological features and prognoses. The main stages of the clonal evolution of SRP, which is already at the early stages and is characterized by pronounced intratumoral genetic heterogeneity, have been determined. However, as PRP progresses, subclones acquire different secondary mutations that contribute to the activation of the same mTOR and VEGF signaling pathways, as well as disrupting the mechanisms of chromatin remodeling and the functioning of TP53. The present program will determine the efficacy of standard doses of axitinib in patients with differentiated mutations in kidney cancer following partial exome sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented metastatic renal cell cancer or cell kidney cancer
* Evidence of measurable disease.
* Adequate renal function (serum creatinine level)
* ECOG Status 0-1
* Patient must provide signed informed consent
* Male or female, age >/= 18 years

Exclusion Criteria:

* Current use or anticipated need for treatment with drugs that are known potent CYP3A4 inhibitors
* Current use or anticipated need for treatment with drugs that are known as potent CYP3A4 or CYP1A2.
* Active gastrointestinal bleeding.
* Severe allergic reactions
* Unwillingness or inability to comply with mandated pretreatment biopsy or therapeutic regimen

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8548775/
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7097956/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/22949125/